CLINICAL TRIAL: NCT03224351
Title: A Phase 2, Randomized, Double-blind, Controlled Study to Evaluate the Safety and Efficacy of VX-659 Combination Therapy in Subjects Aged 18 Years and Older With Cystic Fibrosis
Brief Title: A Study Evaluating the Safety and Efficacy of VX-659 Combination Therapy in Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX16-659-101; 2016-003585-11 (EudraCT Number)
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Results first posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — VX-659; tezacaftor, ivacaftor drug combination; ivacaftor; tezacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1: Placebo (Placebo Comparator): Participants received placebo matched to VX-659/TEZ/IVA in TC treatment period for 4 weeks and placebo matched TEZ/IVA in washout period for 4 days.
  Interventions: Drug: Placebo (matched to VX-659/TEZ/IVA)
- Part 1: VX-659/TEZ/IVA TC - Low Dose (Experimental): Participants received VX-659 80 milligram (mg) once daily (qd)/TEZ 100 mg qd/IVA 150 mg every 12 hours (q12h) in TC treatment period for 4 weeks and TEZ 100 mg qd/IVA 150 mg q12h in washout period for 4 days.
  Interventions: Drug: VX-659; Drug: TEZ/IVA; Drug: IVA
- Part 1: VX-659/TEZ/IVA TC - Medium Dose (Experimental): Participants received VX-659 240 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in TC treatment period for 4 weeks and TEZ 100 mg qd/IVA 150 mg q12h in washout period for 4 days.
  Interventions: Drug: VX-659; Drug: TEZ/IVA; Drug: IVA
- Part 1: VX-659/TEZ/IVA TC - High Dose (Experimental): Participants received VX-659 400 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in TC treatment period for 4 weeks and TEZ 100 mg qd/IVA 150 mg q12h in washout period for 4 days.
  Interventions: Drug: VX-659; Drug: TEZ/IVA; Drug: IVA
- Part 2: TEZ/IVA (Active Comparator): Following run-in period with TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks, participants received TEZ 100 mg qd/IVA 150 mg q12h in TC treatment period for 4 weeks and TEZ 100 mg qd/IVA 150 mg q12h in washout period for 4 weeks.
  Interventions: Drug: TEZ/IVA; Drug: IVA
- Part 2: VX-659/TEZ/IVA TC (Experimental): Following run-in period with TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks, participants received VX-659 400 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in TC treatment period for 4 weeks and TEZ 100 mg qd/IVA 150 mg q12h in washout period for 4 weeks.
  Interventions: Drug: VX-659; Drug: TEZ/IVA; Drug: IVA
- Part 3: Placebo (Placebo Comparator): Participants received placebo matched to VX-659/TEZ/VX-561 in TC treatment period for 4 weeks.
  Interventions: Drug: Placebo (matched to VX-659/TEZ/VX-561)
- Part 3: VX-659/TEZ/VX-561 TC (Experimental): Participants received VX-659 400 mg qd/TEZ 100 mg qd/VX-561 200 mg qd in TC treatment period for 4 weeks.
  Interventions: Drug: VX-659; Drug: TEZ; Drug: VX-561

INTERVENTIONS:
Drug: VX-659 — Tablet for oral administration.
  Arms: Part 1: VX-659/TEZ/IVA TC - High Dose; Part 1: VX-659/TEZ/IVA TC - Low Dose; Part 1: VX-659/TEZ/IVA TC - Medium Dose; Part 2: VX-659/TEZ/IVA TC; Part 3: VX-659/TEZ/VX-561 TC
Drug: TEZ/IVA — TEZ/IVA fixed-dose combination tablet for oral administration.
  Other Names: VX-661/VX-770; Tezacaftor/Ivacaftor
  Arms: Part 1: VX-659/TEZ/IVA TC - High Dose; Part 1: VX-659/TEZ/IVA TC - Low Dose; Part 1: VX-659/TEZ/IVA TC - Medium Dose; Part 2: TEZ/IVA; Part 2: VX-659/TEZ/IVA TC
Drug: IVA — Tablet for oral administration.
  Other Names: VX-770; Ivacaftor
  Arms: Part 1: VX-659/TEZ/IVA TC - High Dose; Part 1: VX-659/TEZ/IVA TC - Low Dose; Part 1: VX-659/TEZ/IVA TC - Medium Dose; Part 2: TEZ/IVA; Part 2: VX-659/TEZ/IVA TC
Drug: Placebo (matched to VX-659/TEZ/IVA) — Placebo matched to VX-659 and TEZ/IVA.
  Arms: Part 1: Placebo
Drug: TEZ — Tablet for oral administration.
  Other Names: VX-661; Tezacaftor
  Arms: Part 3: VX-659/TEZ/VX-561 TC
Drug: VX-561 — Tablet for oral administration.
  Other Names: CTP-656
  Arms: Part 3: VX-659/TEZ/VX-561 TC
Drug: Placebo (matched to VX-659/TEZ/VX-561) — Placebo matched to VX-659, TEZ and VX-561.
  Arms: Part 3: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo- and tezacaftor/ivacaftor (TEZ/IVA)-controlled, parallel-group, 3-part, multicenter study designed to evaluate the safety and efficacy of VX-659 in triple combination (TC) with TEZ and IVA in subjects with cystic fibrosis (CF) who are homozygous for the F508del mutation of the CF transmembrane conductance regulator (CFTR) gene (F/F genotype), or who are heterozygous for the F508del mutation and a minimal function (MF) CFTR mutation not likely to respond to TEZ, IVA, or TEZ/IVA (F/MF genotypes).

ELIGIBILITY:
Key Inclusion Criteria:

* Body weight ≥35 kg.
* Subjects must have an eligibleCFTR genotype.

  * Part 1 and Part 3: Heterozygous for F508del and an MF mutation (F/MF)
  * Part 2: Homozygous for F508del (F/F)
* FEV1 value ≥40% and ≤90% of predicted mean for age, sex, and height

Key Exclusion Criteria:

* History of clinically significant cirrhosis with or without portal hypertension.
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Lung infection with organisms associated with a more rapid decline in pulmonary status.
* History of solid organ or hematological transplantation.

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (47):
- United States (25):
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Miami/Miller School of Medicine, Miami, Florida
  - Advocate Children's Hospital - Park Ridge / North Suburban Pulmonary and Critical Care Consultants, Morton Grove, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - The University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - The Johns Hopkins Hospital/ Johns Hopkins Hospital, David Rubenstein Child Health Building, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Helen DeVos Children's Hospital CF Center, Grand Rapids, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Rutgers-Robert Wood Johnson Medical School/ Rutgers-Robert Wood Johnson Medical School, Clinical Research Center, New Brunswick, New Jersey
  - Albany Medical College, Albany, New York
  - Northwell Health, Long Island Jewish Medical Center, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Respiratory Diseases of Children & Adolescents, Oklahoma City, Oklahoma
  - Children's Hospital of Pittsburgh of University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sanford Research / USD, Sioux Falls, South Dakota
  - University of Tennessee Medical Center-Adult Cystic Fibrosis Clinic, Knoxville, Tennessee
  - Children's Foundation Research Center / Le Bonheur Children's Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah / Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Pediatric Pulmonary & Allergy/Immunology Clinic, Spokane, Washington
- Ireland (4):
  - Cork University Hospital, Cork
  - St. Vincent's University Hosptial, Dublin
  - Galway University Hospitals, Galway
  - University Hospital Limerick, Limerick
- Israel (5):
  - Carmel Medical Center, Haifa
  - Ruth Children's Hospital Rambam Health Care Campus, Haifa
  - Hadassah Medical Organization, Jerusalem
  - The Chaim Sheba medical center, Ramat Gan
  - Schneider Children's Medical Center, Tikvah
- United Kingdom (13):
  - Birmingham Heartlands Hospital, Birmingham
  - Papworth Hospital NHS Foundation Trust, Papworth Everard, Cambridge
  - University Hospital Llandough in Cardiff, Cardiff
  - Royal Devon and Exeter NHS Foundation Trust, Royal Devon and Exeter Hospital, Devon
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, The Royal Victoria Infirmary, Fulham
  - Greater Glasgow and Clyde NHS Board, Glasgow Clinical Research Facility, Glasgow
  - Southampton University Hospitals NHS Foundation Trust, Hampshire
  - Regional Respiratory Centre Belfast City Hospital, London
  - Royal Brompton & Harefied NHS Foundation Trust, London
  - University Hospital of South Manchester NHS Trust, North West Lung Centre, Manchester
  - Liverpool Heart and Chest Hospital, Merseyside
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Ruth Children's Hospital Rambam Health Care Campus, Nottingham

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662
- [Derived] Davies JC, Moskowitz SM, Brown C, Horsley A, Mall MA, McKone EF, Plant BJ, Prais D, Ramsey BW, Taylor-Cousar JL, Tullis E, Uluer A, McKee CM, Robertson S, Shilling RA, Simard C, Van Goor F, Waltz D, Xuan F, Young T, Rowe SM; VX16-659-101 Study Group. VX-659-Tezacaftor-Ivacaftor in Patients with Cystic Fibrosis and One or Two Phe508del Alleles. N Engl J Med. 2018 Oct 25;379(17):1599-1611. doi: 10.1056/NEJMoa1807119. Epub 2018 Oct 18. PMID 30334693

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 124 participants were enrolled in this study (63 in Part 1, 36 in Part 2 and 25 in Part C). Out of 36 participants enrolled in Part 2, 7 participants discontinued treatment in run-in period and were not randomized in triple combination (TC) treatment period. Therefore, below results are presented for 117 participants.
Pre-assignment Details: This study included 3 parts and was conducted in adult participants with cystic fibrosis (CF).
Groups:
- Part 1: Placebo: Participants received placebo matched to VX-659/TEZ/IVA in TC treatment period for 4 weeks and placebo matched to TEZ/IVA in washout period for 4 days.
Period: Overall Study
Arm/Group | Part 1: Placebo | Part 1: VX-659/TEZ/IVA TC - Low Dose | Part 1: VX-659/TEZ/IVA TC - Medium Dose | Part 1: VX-659/TEZ/IVA TC - High Dose | Part 2: TEZ/IVA | Part 2: VX-659/TEZ/IVA TC | Part 3: Placebo | Part 3: VX-659/TEZ/VX-561 TC
Started | 10 | 11 | 20 | 22 | 11 | 18 | 6 | 19
Completed | 10 | 11 | 20 | 22 | 11 | 18 | 6 | 19
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: VX-659/TEZ/IVA TC - Low Dose: Participants received VX-659 80 mg qd/TEZ 100 mg qd/IVA 150 mg every 12 q12h in TC treatment period for 4 weeks and TEZ 100 mg qd/IVA 150 mg q12h in washout period for 4 days.
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo | Part 1: VX-659/TEZ/IVA TC - Low Dose | Part 1: VX-659/TEZ/IVA TC - Medium Dose | Part 1: VX-659/TEZ/IVA TC - High Dose | Part 2: TEZ/IVA | Part 2: VX-659/TEZ/IVA TC | Part 3: Placebo | Part 3: VX-659/TEZ/VX-561 TC | Total
Number analyzed (Participants) | 10 | 11 | 20 | 22 | 11 | 18 | 6 | 19 | 117
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=18 and <65 years | 10 | 11 | 20 | 22 | 11 | 18 | 6 | 19 | 117
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 7 | 12 | 4 | 6 | 3 | 11 | 54
  Male | 6 | 4 | 13 | 10 | 7 | 12 | 3 | 8 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 6
  Not Hispanic or Latino | 10 | 11 | 18 | 22 | 10 | 17 | 5 | 18 | 111
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  White | 10 | 11 | 20 | 22 | 11 | 16 | 6 | 17 | 113
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) [Count of Participants; unit: Participants] — FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
  Participants
    <40 percent | 2 | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 8
    ≥40 to <70 percent | 6 | 9 | 13 | 13 | 8 | 12 | 5 | 13 | 79
    ≥70 to ≤90 percent | 2 | 2 | 6 | 7 | 3 | 5 | 1 | 4 | 30
    >90 percent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 Through Safety Follow-up (up to Day 61 for Part 1, Day 85 for Part 2 and Day 57 for Part 3)
Population: Safety Set included all participants who received at least 1 dose of study drug in TC treatment period.
Measure: Number; unit: participants
Arm/Group | Part 1: Placebo | Part 1: VX-659/TEZ/IVA TC - Low Dose | Part 1: VX-659/TEZ/IVA TC - Medium Dose | Part 1: VX-659/TEZ/IVA TC - High Dose | Part 2: TEZ/IVA | Part 2: VX-659/TEZ/IVA TC | Part 3: Placebo | Part 3: VX-659/TEZ/VX-561 TC
Number analyzed (Participants) | 10 | 11 | 20 | 22 | 11 | 18 | 6 | 19
participants
  Participants with TEAEs | 9 | 10 | 15 | 17 | 9 | 15 | 6 | 18
  Participants with SAEs | 3 | 1 | 4 | 1 | 2 | 1 | 3 | 2

2. Primary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline Through Day 29
Population: Full Analysis Set (FAS) included all randomized participants with an eligible cystic fibrosis transmembrane conductance regulator protein (CFTR) genotype and received at least 1 dose of study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage points
Groups:
- Part 2: TEZ/IVA: Following run-in period with TEZ 100 mg qd/IVA 150 mg q12h for 4 weeks, participants TEZ 100 mg qd/IVA 150 mg q12h in TC treatment period for 4 weeks and TEZ 100 mg qd/IVA 150 mg q12h in washout period for 4 weeks.
Arm/Group | Part 1: Placebo | Part 1: VX-659/TEZ/IVA TC - Low Dose | Part 1: VX-659/TEZ/IVA TC - Medium Dose | Part 1: VX-659/TEZ/IVA TC - High Dose | Part 2: TEZ/IVA | Part 2: VX-659/TEZ/IVA TC | Part 3: Placebo | Part 3: VX-659/TEZ/VX-561 TC
Number analyzed (Participants) | 10 | 11 | 20 | 22 | 11 | 18 | 6 | 19
percentage points | 0.4 [-5.3 to 6.1] | 10.2 [4.8 to 15.5] | 12.0 [8.0 to 16.0] | 13.3 [9.5 to 17.1] | 0.0 [-3.9 to 3.9] | 9.7 [6.6 to 12.7] | -5.0 [-12.2 to 2.1] | 12.2 [8.3 to 16.2]

3. Secondary Outcome: Absolute Change in Sweat Chloride Concentrations
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline Through Day 29
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Arm/Group | Part 1: Placebo | Part 1: VX-659/TEZ/IVA TC - Low Dose | Part 1: VX-659/TEZ/IVA TC - Medium Dose | Part 1: VX-659/TEZ/IVA TC - High Dose | Part 2: TEZ/IVA | Part 2: VX-659/TEZ/IVA TC | Part 3: Placebo | Part 3: VX-659/TEZ/VX-561 TC
Number analyzed (Participants) | 10 | 11 | 20 | 22 | 11 | 18 | 6 | 19
millimole per liter (mmol/L) | 2.9 [-6.3 to 12.2] | -45.7 [-54.4 to -37.0] | -43.8 [-50.7 to -37.0] | -51.4 [-57.8 to -44.9] | 3.0 [-2.8 to 8.9] | -42.2 [-46.8 to -37.7] | -1.3 [-12.4 to 9.8] | -38.1 [-44.4 to -31.8]

4. Secondary Outcome: Relative Change in ppFEV1
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline Through Day 29
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Part 1: Placebo | Part 1: VX-659/TEZ/IVA TC - Low Dose | Part 1: VX-659/TEZ/IVA TC - Medium Dose | Part 1: VX-659/TEZ/IVA TC - High Dose | Part 2: TEZ/IVA | Part 2: VX-659/TEZ/IVA TC | Part 3: Placebo | Part 3: VX-659/TEZ/VX-561 TC
Number analyzed (Participants) | 10 | 11 | 20 | 22 | 11 | 18 | 6 | 19
percent change | 0.0 [-10.5 to 10.4] | 18.8 [8.9 to 28.7] | 21.1 [13.8 to 28.5] | 24.6 [17.6 to 31.6] | 0.1 [-7.1 to 7.3] | 17.3 [11.7 to 23.0] | -11.3 [-23.7 to 1.1] | 21.5 [14.6 to 28.4]

5. Secondary Outcome: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: From Baseline at Day 29
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Part 1: VX-659/TEZ/IVA TC - High Dose: Participants received VX-659 400 mg qd/TEZ 100 mg/IVA 150 mg q12h in TC treatment period for 4 weeks and TEZ 100 mg qd/IVA 150 mg q12h in washout period for 4 days.
Arm/Group | Part 1: Placebo | Part 1: VX-659/TEZ/IVA TC - Low Dose | Part 1: VX-659/TEZ/IVA TC - Medium Dose | Part 1: VX-659/TEZ/IVA TC - High Dose | Part 2: TEZ/IVA | Part 2: VX-659/TEZ/IVA TC | Part 3: Placebo | Part 3: VX-659/TEZ/VX-561 TC
Number analyzed (Participants) | 10 | 11 | 20 | 22 | 11 | 18 | 6 | 19
units on a scale | 4.7 [-7.5 to 16.8] | 24.6 [13.0 to 36.2] | 19.8 [11.0 to 28.6] | 21.8 [13.6 to 30.0] | 2.9 [-5.2 to 11.1] | 19.5 [13.1 to 25.9] | -4.1 [-17.8 to 9.6] | 14.7 [7.1 to 22.4]

6. Secondary Outcome: Observed Pre-dose Concentration (Ctrough) of VX-659, TEZ, M1-TEZ, IVA, M1-IVA, and VX-561
Time Frame: Pre-dose at Day 15 and Day 29
Population: Pharmacokinetic Set (PK) included all participants who have received at least 1 dose of study drug in TC treatment period. Here "Number Analyzed" signifies those participants who were evaluable at specified time points. VX-659 category was not applicable for Part 2: TEZ/IVA group. VX-561 category was applicable for Part 3: TC group only. IVA and M1-IVA categories were not applicable for Part 3: TC group.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1: VX-659/TEZ/IVA TC - Low Dose | Part 1: VX-659/TEZ/IVA TC - Medium Dose | Part 1: VX-659/TEZ/IVA TC - High Dose | Part 2: TEZ/IVA | Part 2: VX-659/TEZ/IVA TC | Part 3: VX-659/TEZ/VX-561 TC
Number analyzed (Participants) | 11 | 20 | 22 | 11 | 18 | 19
nanogram per milliliter (ng/mL)
  VX-659: Day 15: number analyzed (Participants) | 10 | 16 | 19 | 0 | 17 | 17
  VX-659: Day 15 | 393 (604) | 622 (429) | 1100 (731) |  | 835 (474) | 1140 (646)
  VX-659: Day 29: number analyzed (Participants) | 11 | 19 | 22 | 0 | 18 | 19
  VX-659: Day 29 | 566 (861) | 699 (489) | 1080 (582) |  | 1070 (914) | 923 (582)
  TEZ: Day 15: number analyzed (Participants) | 10 | 16 | 19 | 7 | 17 | 17
  TEZ: Day 15 | 1910 (1360) | 1250 (907) | 1110 (455) | 1050 (473) | 1350 (1440) | 1000 (305)
  TEZ: Day 29: number analyzed (Participants) | 11 | 19 | 22 | 11 | 18 | 19
  TEZ: Day 29 | 1910 (1230) | 1050 (553) | 1010 (479) | 1150 (480) | 955 (422) | 776 (321)
  M1-TEZ: Day 15: number analyzed (Participants) | 10 | 16 | 19 | 7 | 17 | 19
  M1-TEZ: Day 15 | 4390 (949) | 3710 (1230) | 4280 (1190) | 4160 (1260) | 4010 (1210) | 4060 (660)
  M1-TEZ: Day 29: number analyzed (Participants) | 11 | 19 | 22 | 11 | 18 | 19
  M1-TEZ: Day 29 | 4300 (774) | 3650 (1280) | 3870 (1020) | 3790 (1080) | 3810 (1120) | 3660 (1190)
  IVA: Day 15: number analyzed (Participants) | 10 | 16 | 19 | 7 | 17 | 0
  IVA: Day 15 | 824 (781) | 522 (567) | 423 (261) | 458 (239) | 313 (158) |
  IVA: Day 29: number analyzed (Participants) | 11 | 19 | 22 | 11 | 18 | 0
  IVA: Day 29 | 719 (604) | 443 (398) | 371 (220) | 490 (179) | 296 (175) |
  M1-IVA: Day 15: number analyzed (Participants) | 10 | 16 | 19 | 7 | 17 | 0
  M1-IVA: Day 15 | 1200 (711) | 1050 (852) | 1170 (674) | 1310 (684) | 844 (622) |
  M1-IVA Day 29: number analyzed (Participants) | 11 | 19 | 22 | 11 | 18 | 0
  M1-IVA Day 29 | 1130 (682) | 1140 (950) | 1030 (460) | 1240 (321) | 866 (691) |
  VX-561: Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 17
  VX-561: Day 15 |  |  |  |  |  | 380 (240)
  VX-561: Day 29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 19
  VX-561: Day 29 |  |  |  |  |  | 288 (165)

ADVERSE EVENTS:
Time Frame: Day 1 Through Safety Follow-up (up to Day 61 for Part 1, Day 85 for Part 2 and Day 57 for Part 3)
Arm/Group | Part 1: Placebo | Part 1: VX-659/TEZ/IVA TC - Low Dose | Part 1: VX-659/TEZ/IVA TC - Medium Dose | Part 1: VX-659/TEZ/IVA TC - High Dose | Part 2: TEZ/IVA | Part 2: VX-659/TEZ/IVA TC | Part 3: Placebo | Part 3: VX-659/TEZ/VX-561 TC
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11 | 0/20 | 0/22 | 0/11 | 0/18 | 0/6 | 0/19
Serious Adverse Events (participants affected / at risk) | 3/10 | 1/11 | 4/20 | 1/22 | 2/11 | 1/18 | 3/6 | 2/19
Other Adverse Events (participants affected / at risk) | 8/10 | 10/11 | 15/20 | 17/22 | 8/11 | 15/18 | 5/6 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=10) | Part 1: VX-659/TEZ/IVA TC - Low Dose (N=11) | Part 1: VX-659/TEZ/IVA TC - Medium Dose (N=20) | Part 1: VX-659/TEZ/IVA TC - High Dose (N=22) | Part 2: TEZ/IVA (N=11) | Part 2: VX-659/TEZ/IVA TC (N=18) | Part 3: Placebo (N=6) | Part 3: VX-659/TEZ/VX-561 TC (N=19)
Pulmonary function test decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2 | 1 | 2 | 1 | 2 | 1 | 3 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=10) | Part 1: VX-659/TEZ/IVA TC - Low Dose (N=11) | Part 1: VX-659/TEZ/IVA TC - Medium Dose (N=20) | Part 1: VX-659/TEZ/IVA TC - High Dose (N=22) | Part 2: TEZ/IVA (N=11) | Part 2: VX-659/TEZ/IVA TC (N=18) | Part 3: Placebo (N=6) | Part 3: VX-659/TEZ/VX-561 TC (N=19)
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 3
Fatigue (General disorders) | 0 | 2 | 2 | 0 | 1 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Application site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exercise tolerance decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1 | 3 | 2 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Bacterial test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Weight increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pulmonary function test decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood glucose fluctuation (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coronavirus test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Crystal urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Forced expiratory volume decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glucose urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Monocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Red blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary sediment present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 6 | 4 | 2 | 4 | 2 | 4
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 3 | 1 | 3 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 4 | 0 | 2 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 4 | 4 | 0 | 3 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 2 | 2 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatic failure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 2 | 1 | 3 | 1 | 4 | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1 | 3 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Genital infection fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT03224351/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT03224351/SAP_001.pdf